CLINICAL TRIAL: NCT06684444
Title: Assessing Clinical Effectiveness and Implementation of Worksite Sleep Health Coaching in Firefighters
Brief Title: Evaluating Worksite Sleep Health Coaching in Firefighters: The Sleep Assistance for Firefighters Study
Acronym: SAFFIRE
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001612; R01HL162799 (NIH)
Record Dates: First submitted 2024-10-31; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Behavioral Therapy; Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Sleep Disorders, Intrinsic
Keywords: CBTi; sleep deprivation; sleep disorders; firefighters; sleep health coaching
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Sleep Disorders, Intrinsic; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (firefighter Sleep Health Coaching Intervention [ffSHC]) (Experimental): In this arm, fire service employees receive a structured sleep health intervention based on Cognitive Behavioral Therapy for Insomnia (CBTi). The intervention includes sleep health promotion, telephone-administered sleep coaching, and implementation strategies to promote better sleep practices. Each cluster will transition from the control arm to this intervention at a fixed time, and outcome data will be collected at multiple time points during and after the intervention phase to assess its effectiveness.
  Interventions: Behavioral: firefighter Sleep Health Coaching Intervention (ffSHC)
- Control (Minimally Enhanced Usual Care) (Active Comparator): In this arm, fire service workers receive usual care with minimal enhancements but without the full sleep health intervention. During this phase, clusters will serve as the control group, and data on sleep health and related outcomes will be collected for comparison against the intervention phase. Each cluster will remain in this arm until a predetermined time point, at which they transition to the intervention arm after a one-month preparation phase.
  Interventions: Behavioral: Control (Minimally Enhanced Usual Care)

INTERVENTIONS:
Behavioral: firefighter Sleep Health Coaching Intervention (ffSHC) — This multi-component intervention is based on principles of cognitive behavioral therapy for insomnia. It includes telephone-based sleep health coaching to individuals, targeted training and sleep health education to fire service leaders, agency-level sleep health promotion, and facilitation strategies to internal facilitators.
  Arms: Intervention (firefighter Sleep Health Coaching Intervention [ffSHC])
Behavioral: Control (Minimally Enhanced Usual Care) — The control arm is minimally enhanced usual care. Usual care interventions for sleep disturbance include any health or wellness interventions administered by the agency on the topic of sleep, including occupational health intervention, employee assistance programs, education, signage, and webinars. The type and dose of care will be assessed at each timepoint. Minimal enhancement is a referral to the agency's Employee Assistance Program and will address the ethical problem in the control condition of identifying but not treating a sleep disturbance.
  Arms: Control (Minimally Enhanced Usual Care)

SUMMARY:
Insufficient sleep is a significant public health issue, particularly affecting shift workers like firefighters, nearly half of whom report short or poor-quality sleep, with 35-40% screening positive for sleep disorders. Cognitive Behavioral Therapy for Insomnia (CBTi) is a recommended and effective treatment, but access to such interventions remains low. This study will recruit 20 fire agencies in Arizona (400 firefighters) to test if a CBTi-informed intervention, including sleep health coaching and agency-wide promotion, improves sleep more effectively than usual care. The trial will also explore factors that influence successful implementation across agencies.

DETAILED DESCRIPTION:
Insufficient sleep is a major public health crisis in the United States and worldwide, disproportionately affecting shift workers and other at-risk groups. Firefighters are one such group at heightened risk for disturbed sleep. Almost half of career firefighters report short sleep and poor sleep quality, and 35-40% of firefighters screen positive for a sleep disorder.

Evidence-based sleep health interventions are available and highly effective in eliciting behavioral change. The American College of Physicians recommends Cognitive Behavioral Therapy for Insomnia (CBTi) as the first-line treatment for Insomnia Disorder, and substantial evidence supports the efficacy of this therapy with comorbid conditions, including shiftwork and obstructive sleep apnea. Unfortunately, access to CBT-informed sleep health interventions remains low. Workplace wellness programs could be one way to help more firefighters receive sleep intervention.

This study will recruit 20 fire agencies in Arizona (n = 400 career firefighters) to examine whether a CBTi-informed intervention is more effective than usual care in reducing sleep disturbances or improving multidimensional sleep health. The intervention will last one year and will include telephone-administered sleep health coaching to firefighters, sleep health promotion to the agency and agency leaders, and external/internal facilitation strategies for implementation. The trial will also examine which combinations of factors are associated with successful agency implementation of the intervention. All participating agencies will receive the intervention; however, some agencies will wait longer to receive the intervention than others.

ELIGIBILITY:
Inclusion Criteria:

* Required to be employed as career (paid), uniformed fire service workers that must work in a participating fire agency.
* Must have moderate or more severe levels of sleep disturbances [item-level calibrated T-score of 55 or higher on the 8-item Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SD) questionnaire].
* Must have private access to a computer or phone for sleep health coaching.

Exclusion Criteria:

* Children younger than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Disturbance questionnaire | 6 assessments, 6 months apart
  PROMIS measures are scored on the T-score metric. 50 is the mean score of a relevant reference population, and 10 is the standard deviation of that population. High scores mean more of the concept being measured.
Multidimensional sleep health (MSH) composite | 6 assessments, 6 months apart
  The composite uses weighted summaries of the z-scores of four actigraphic sleep health dimensions: regularity, timing, sleep efficacy, sleep duration and two subjective sleep health dimensions: satisfaction and alertness, derived from items on the PROMIS-SD and PROMIS Sleep Related Impairment (PROMIS-SRI) scale respectively. High scores mean less of the concept being measured (i.e., worse sleep health).

SECONDARY OUTCOMES:
PROMIS Sleep Related Impairment questionnaire | 6 assessments, 6 months apart
  PROMIS measures are scored on the T-score metric. 50 is the mean score of a relevant reference population, and 10 is the standard deviation of that population. High scores mean more of the concept being measured.
Wake time after sleep onset (WASO), min - actigraphy | 6 assessments, 6 months apart
  This index derived from wrist-worn actigraphy provides an average estimate of the total number of minutes awake after initial sleep onset. High scores mean more of the concept being measured.
Number of awakenings (NAW) - actigraphy | 6 assessments, 6 months apart
  This index derived from wrist-worn actigraphy provides an average estimate of the total number of awakenings or arousals during the sleep period. High scores mean more of the concept being measured.

OTHER OUTCOMES:
Blood pressure | 6 assessments, 6 months apart
  Systolic and diastolic blood pressure (mm Hg)
Heart rate | 6 assessments, 6 months apart
  Nocturnal heart rate, difference between mean nocturnal and daytime heart rate
Occupational health clinic assessments-1, CVD | 4 assessments, approximately 1 year apart
  cholesterol
Occupational health clinic assessments-2, CVD | 4 assessments, approximately 1 year apart
  body mass index (BMI)
Occupational health clinic assessments-3, CVD | 4 assessments, approximately 1 year apart
  blood pressure (mm Hg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets will be stripped of personally identifiable information (PII) data elements. IPD shared include: intervention condition, data from surveys and interviews, and individual-level summaries of actigraphic indices, heart rate, and blood pressure data collected across six timepoints (3 years). Survey responses related to sensitive information will not be shared.
Time Frame: Data will be made available on National Sleep Research Resource (NSRR) repository to other users no later than the time of an associated publication or at the end of the performance period, whichever comes first. Primary data will be available for a minimum of 10 years after the end of the performance period, consistent with University of Arizona policy.
Access Criteria: Access to the resources at NSRR is controlled by per-dataset-access control, and access is only granted to individuals who have completed the web-based Data Access and Use Agreement (DAUA). Each DAUA submission is reviewed by the NSRR Review Committee, and reviewers ascertain that use of data appears appropriate with the intention of data collected and that there is a commitment to keep the data stored securely by the end-user. NSRR DAUAs expire 3 years from the date access is granted and can be renewed by either submitting a new request for data access or by requesting an extension of the agreement in writing to the NSRR Review Committee.
URL: https://sleepdata.org/